CLINICAL TRIAL: NCT00044707
Title: Evaluation of an Orally Administered Medication When Taken in Conjunction With Pramlintide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 137-154
Record Dates: First submitted 2002-09-03; First posted 2002-09-05 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — pramlintide

ARMS (2):
- Pramlintide acetate (AC137) (Active Comparator): Pramlintide acetate (AC137) injection is a clear, colorless, sterile solution for SC injection. It consists of pramlintide in sodium acetate buffer, pH 4.0, containing 43 mg/mL mannitol as an iso-osmolality modifier and 2.25 mg/mL metacresol as a preservative. The strength of pramlintide injection is 0.6 mg/mL
  Interventions: Drug: Pramlintide acetate
- Placebo (Placebo Comparator): Placebo solution is the same, sterile preserved formulation, except the active ingredient, pramlintide, is omitted

INTERVENTIONS:
Drug: Pramlintide acetate — Clear, colorless, sterile solution for SC injection.
  Arms: Pramlintide acetate (AC137)

SUMMARY:
This is a randomized, single-blind, placebo-controlled, crossover study to examine the effect of pramlintide on the pharmacokinetics of an orally administered medication

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus treated with diet and/or oral agents
* HbA1c 6.5-11.0

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2002-08; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
To determine the effect of pramlintide on the PK of an oral medication | 7 Days
  To determine the effect of pramlintide on the pharmacokinetics of an orally administered concomitant medication (acetaminophen) when administered at various times in relation to subcutaneous (SC) pramlintide dosing. The noncompartmental plasma acetaminophen pharmacokinetic (PK) parameters used in the analyses are defined as follows: AUC(0-12hr): Area under the plasma acetaminophen concentration-time curve. Cmax : The peak acetaminophen concentrationd. Tmax : Duration from the time of acetaminophen dosing to the time of the first maximum observed concentration, Cmax.
  t½: Terminal half-life
  The primary study endpoints include:
  * pharmacokinetic parameters AUC(0-12 hr) and Cmax of plasma acetaminophen concentrations Secondary Study Endpoints
  * pharmacokinetic parameters Tmax and t1/2 of plasma acetaminophen concentrations

SECONDARY OUTCOMES:
safety and tolerability as measured by analysis of laboratory values and adverse events | 7 Days
  To assess safety and tolerability of pramlintide SC injection, including adverse events, as a function of the timing of an orally administered concomitant medication (acetaminophen).

CONTACTS AND LOCATIONS:
Locations (1):
- ICSL-Clinical Studies, Fort Lauderdale, Florida, United States